CLINICAL TRIAL: NCT03449004
Title: The Online Patient Satisfaction Index (OPSI): Development and Validation Among Patients With Low Back Pain
Brief Title: Development and Validation of the Online Patient Satisfaction Index
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Allan Riis, Senior researcher, Aalborg University Hospital
Other Study IDs: AllanRiis_10; TamanaAfzali (Other: Aalborg University)
Record Dates: First submitted 2018-02-14; First posted 2018-02-28 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Low Back Pain
Keywords: Validation; questionnaire; satisfaction; online information
MeSH Terms: conditions — Low Back Pain; Personal Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Validation of the OPSI questionnaire — A questionnaire to measure satisfaction with online information for patients with low back pain
  Other Names: The Online Patient Satisfaction Index

SUMMARY:
Low Back Pain (LBP) is the most common musculoskeletal disorder and a leading cause of disability worldwide. It is the most frequent reason for consulting general practice and has an impact on daily life and work capacity. A cornerstone in treating LBP is the provision of information to patients, and the internet is increasingly being used as a source of health information delivery. However, the effect of and satisfaction with online information have been questioned. The investigators aimed to develop and validate a multi-item instrument to measure an index score of satisfaction of online information for patients with LBP.

The conceptualization of a Patient Reported Outcome (PRO) to measure a multidimensional index score is modelled on the assumption of a causal relationship between domains of experiences with online information and patients' combined index score of satisfaction. Findings from 15 patient interviews was applied to draft the first version of the instrument. Followed by pilot testing on patients (n=20) and experts (n=7) before validating the instrument on patients (n=150). Patients were eligible for inclusion if they had their first onset of LBP for 14 days. Patients were included regardless of pain intensity. Patients were excluded if they did not have Internet access, were pregnant, did not speak Danish as their native language, or had signs of serious underlying disease.

DETAILED DESCRIPTION:
BACKGROUND Low back pain (LBP) is highly prevalent and a frequent reason for patients to consult general practice. It is a common pain condition affecting both men and women at all ages. LBP is rarely caused by only one specific factor but is eventually caused by multiple and often unknown factors. This makes it difficult to perform a precise diagnosis based on a single cause and for most patients, the LBP is diagnosed as nonspecific with or without nerve root compression.

Patient education and information is a cornerstone in the management of LBP. Providing information to patients is considered a crucial issue as it is necessary to support self-management. However, the delivery of evidence based information by a healthcare professional is time consuming and not straight forward to deliver during the available consultation time in general practice.

The internet is a widely accessible source of medical information to patients and offer a range of information provided by a variety of different sources. It has been reported that about 50% of patients use internet search for health and medical advice, and evidence suggests that patients willingness to use this source to obtain information about their health is increasing. The advance of new technologies offer new opportunities to the delivery of patient information on private computers, tablets, and smartphones. Online information can be considered an inexpensive solution to extend the combined treatment in general practice. Therefore, future optimization of information delivery has the potential to increase the delivery of evidence-based treatment of LBP which may lead to better patient outcomes. Patient satisfaction has been suggested as an important domain when evaluating the provision of online information.

Measuring patient satisfaction is a recommended outcome measure when evaluating the effect of interventions for LBP. Furthermore, patient satisfaction may be associated with compliance to the recommended treatment. Patient satisfaction is, however, rarely applied as the primary outcome in studies of LBP. To the investigators' knowledge, there exist no instrument to evaluate specific satisfaction with information delivered online for LBP. The aim of this study is to develop and validate a new questionnaire to inform about patients' satisfaction with online information for LBP.

METHODS This is a development and validation study of a patient reported questionnaire to (1) inform about the discrepancy in satisfaction of online information for LBP between groups and (2) to evaluate changes in satisfaction over time. The conceptualization is based on a formative model, which assumes a causal relationship between different domains of satisfaction with online information and the construct of patients' combined index score of satisfaction. The first version of the instrument was based on findings from an interview study among patients consulting for LBP in Danish general practice. Data for further developing on the first version were exclusively collected for piloting and validating the instrument.

HYPOTHESIS The OPSI index scores among patients categorised as promoters will be compared to the OPSI index scores of patients categorised as non-promotors on the Net Promotor Score. Based on results from the pilot test. It is hypothesised that promotors will have an OPSI score of minimum 2.5 points more than non-promotors (0-8 Points on the Net Promotor Score).

ELIGIBILITY:
Inclusion Criteria:

During the last year experienced LBP of any pain intensity. Regardless of present pain at inclusion.

Exclusion Criteria:

* no internet access
* pregnant women
* not able to speak/read Danish
* spinal stenosis
* serious underlying disease for low back pain (e.g. signs of fracture, cauda equina syndrome, malignancy, osteoporosis, or spondyloarthritis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with low back pain during the last year. Patients are recruited from social media and The SANO centre, a rehabilitation center for patients with musculoskeletal pain conditions. If recruitment will be difficult we will combine with recruitment from poster in waiting rooms at primary care physicians, physiotherapists, and/or chiropractors.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Association between the Online Patient Satisfaction Index (0-24 Points, higher scores indicate higher satisfaction) and the Net Promotor Score (10-0 Points, 10-9 Points is categorised as promotors and 8-0 Points is categorised as non-promotors) | Cross sectional (< 45 seconds)
  Convergent validity

SECONDARY OUTCOMES:
Association between the Online Patient Satisfaction Index (0-24 Points, higher score is indicating higher satisfaction) and the Roland Morris Disability questionnaire (RMDQ, 0-23 Points, a high score is indicating high disability) | Cross sectional (< 45 seconds)
  Discriminant validity
Test re-test of the Online Patient Satisfaction Index (0-24 Points, higher score is indicating higher satisfaction) | One week
  Reliability (subpopulation of 50 patients)
Association between the Online Patient Satisfaction Index (0-24 Points, higher scores indicate higher satisfaction) and global rating of satisfaction (10-0 Points, 10-9 Points is categorised as satisfied and 8-0 Points is categorised as not satisfied) | Cross sectional (< 45 seconds)
  Convergent validity

CONTACTS AND LOCATIONS:
Overall Officials: Janus L Thomsen, PhD, Study Chair — Research unit for General Practice in Aalborg, Denmark
Locations (1):
- Research Unit for General Practice in Aalborg, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kent PM, Keating JL. The epidemiology of low back pain in primary care. Chiropr Osteopat. 2005 Jul 26;13:13. doi: 10.1186/1746-1340-13-13. PMID 16045795
- [Background] Croft PR, Macfarlane GJ, Papageorgiou AC, Thomas E, Silman AJ. Outcome of low back pain in general practice: a prospective study. BMJ. 1998 May 2;316(7141):1356-9. doi: 10.1136/bmj.316.7141.1356. PMID 9563990
- [Background] Hoy D, Brooks P, Blyth F, Buchbinder R. The Epidemiology of low back pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):769-81. doi: 10.1016/j.berh.2010.10.002. PMID 21665125
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] National Guideline Centre (UK). Low Back Pain and Sciatica in Over 16s: Assessment and Management. London: National Institute for Health and Care Excellence (NICE); 2016 Nov. Available from http://www.ncbi.nlm.nih.gov/books/NBK401577/ PMID 27929617
- [Background] Diaz JA, Griffith RA, Ng JJ, Reinert SE, Friedmann PD, Moulton AW. Patients' use of the Internet for medical information. J Gen Intern Med. 2002 Mar;17(3):180-5. doi: 10.1046/j.1525-1497.2002.10603.x. PMID 11929503
- [Background] Tustin N. The role of patient satisfaction in online health information seeking. J Health Commun. 2010 Jan;15(1):3-17. doi: 10.1080/10810730903465491. PMID 20390974
- [Background] A. Riis, M. B. Jensen, A. M. Kanstrup, J. Hartvigsen, M. S. Rathleff, D. M. Hjelmager, L. D. Vinther, and P. Bertelsen, "Tailored on-line information and advice to patients with low back pain in general practice," 2016.
- [Background] Deyo RA, Diehl AK. Patient satisfaction with medical care for low-back pain. Spine (Phila Pa 1976). 1986 Jan-Feb;11(1):28-30. doi: 10.1097/00007632-198601000-00008. PMID 2939566
- [Derived] Afzali T, Lauridsen HH, Thomsen JL, Hartvigsen J, Jensen MB, Riis A. The Online Patient Satisfaction Index for Patients With Low Back Pain: Development, Reliability, and Validation Study. JMIR Form Res. 2021 Nov 15;5(11):e21462. doi: 10.2196/21462. PMID 34779785